CLINICAL TRIAL: NCT05201573
Title: DIAM™ Spinal Stabilization System Long Term Follow up Clinical Plan
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Companion Spine, LLC (Other)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Other Study IDs: CP21001
Record Dates: First submitted 2022-01-06; First posted 2022-01-21 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain | interventions — Watchful Waiting

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Subjects historically treated with DIAM: Subjects randomized to the DIAM arm and treated with the DIAM™ Spinal Stabilization System in the IDE study OR randomized to the Control arm and crossed over to receive treatment with the DIAM™ Spinal Stabilization System in the IDE study
  Interventions: Other: Observational

INTERVENTIONS:
Other: Observational — This is an observational study of long term follow up data for patients who previously received the DIAM implant

SUMMARY:
A hybrid prospective/retrospective, multicenter, single-arm, data collection study.

DETAILED DESCRIPTION:
Collect long-term follow-up data with x-rays and CT on subjects who received the DIAM™ Spinal Stabilization System through the original IDE protocol.

Data collected at one-time point from subjects with at least 5 years of follow-up data.

ELIGIBILITY:
Inclusion Criteria:

* Subject randomized to the DIAM arm and treated with the DIAM™Spinal Stabilization System in the IDE study OR randomized to the Control arm and crossed over to receive treatment with the DIAM™ Spinal Stabilization System in the IDE study.
* Willing and able to consent to study procedures

Exclusion Criteria:

* NA

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data will be collected from up to 8 sites that participated in the DIAM Pivotal Study.
  There is no randomization for this study. The goal is to collect long-term follow-up data on patients who participated in the DIAM™Spinal Stabilization System - Pivotal Study and were randomized to the DIAM arm or who were randomized to the control arm AND crossed over to receive DIAM treatment.
Sampling Method: Non-Probability Sample
Enrollment: 175 (Estimated)
Dates: Start 2022-01-17 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety associated with the use of the investigational implant during long term follow up | 5-10 years after implantation
  The DIAM device, specifically at long-term follow-up. A subject is considered to be a long-term success if they are free from serious device-related adverse events through final follow-up.
  Secondary surgical intervention for treatment failure (i.e. recurrence of pain or functional impairment) without other serious device-related adverse event is not considered to be a serious device-related adverse event for the purposes of the primary endpoint.

SECONDARY OUTCOMES:
Back Pain evaluation | 5-10 years after implantation
  Composite overall success consisting of:
  Pain/disability (Oswestry) success (≥15 pt. improvement relative to baseline) No serious adverse event is classified as "implant-associated", "procedure associated" or "implant-/surgical procedure associated." No additional surgical procedure at the involved level is classified as a failure.
Back Pain evaluation | 5-10 years after implantation
  Change in back pain score compared to baseline
Back Pain evaluation | 5-10 years after implantation
  Back pain success calculated as: Pre-treatment Score - Post-treatment Score > 0 (Score = pain intensity + pain frequency)
Back Pain evaluation | 5-10 years after implantation
  SF-36/RAND-36 success calculated by: PCSPost-tx - PCSPre-tx > 0

IPD SHARING:
Plan to Share IPD: Undecided